CLINICAL TRIAL: NCT05134792
Title: Effect of Pre-emptive Intravenous Immunoglobulin Administration on the Incidence of Septic Episodes in Pediatric Burn Patients: A Randomized Controlled Study
Brief Title: Effect of Pre-emptive Intravenous Immunoglobulin (IVIG) on the Incidence of Septic Episodes in Pediatric Burn Patients
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Hanan Mostafa ,MD, Lecturer of Anesthesia ,surgical intensive care and Pain ., Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Pt 2221
Record Dates: First submitted 2021-11-02; First posted 2021-11-26 (Actual); Last update posted 2022-11-15 (Actual); Status verified 2022-11

CONDITIONS: Burn Shock
MeSH Terms: interventions — Immunoglobulins, Intravenous

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- No intravenous immunoglobulin (IVIG) (No Intervention): The control group are burn patients with inclusion criteria that did not receive IVIG.
- Intravenous immunoglobulin (IVIG) group (Experimental): Pediatric burn patients between 1and 5 years with 10% or greater burn area of TBSA within 24 hours of onset of burn will receive intravenous immunoglobulin.
  Interventions: Drug: intravenous immunoglobulin

INTERVENTIONS:
Drug: intravenous immunoglobulin — All pediatric burn patients allocated in group intra venous immunoglobulin admitted will receive 200 mg/kg IVIG once after their initial resuscitation before 48 hours passes of burn incident.
  Other Names: LIV GAMMA "S/D treated Human Immunoglobulin "2.5 grams/50 ml
  Arms: Intravenous immunoglobulin (IVIG) group

SUMMARY:
Effect of pre-emptive intravenous immunoglobulin administration on the incidence of septic episodes in pediatric burn patients: A randomized controlled study.

DETAILED DESCRIPTION:
After randomization, Treatment and control groups will receive Parkland formula (4 ml/kg per percent total burn surface area; (TBSA), counting moderate (partial thickness) and severe (full thickness) burn area only) using Ringer's lactate solution (half of the fluid will be given over the first eight hours and the remaining half will be given over the next 16 hours), plus normal 24-hour maintenance fluid requirements using glucose solution.

When initiating Parkland, treatment group (Group A) will receive intravenous immunoglobulin IVIG (LIV-GAMMA "S/D treated Human Immunoglobulin" 2.5 grams/50 ml) with a dose of 200 mg/kg once on admission.

* On each septic or septic shock episode in either groups, the patients will be treated with appropriate antibiotics empirically or culture-based.

  * Assessments
  * On admission, all patients included in the study will be fully examined clinically to identify the extent and area of burn and clinical signs of infection or dehydration as fever, respiratory rate, urinary output and capillary refill. Besides, non-invasive blood pressure (systolic blood pressure (SBP), diastolic blood pressure (DBP) and mean arterial blood pressure (MAP)), electrocardiogram and arterial oxygen saturation will be assessed.
  * Parameters to be measured
* Serum immunoglobulin G( IgG) level,
* Serum micro RNA (miR-25) ,
* Serum C reactive protein (CRP) level,
* Serum lactate,
* Serum Procalcitonin
* Serum Malondialdehyde(MDA).
* Serum Glutathione Peroxidase .

  * In addition, Complete Blood picture with differential, coagulation profile, liver function tests (alanine transaminase (ALT), aspartate amino transferase(AST), Albumin and Bilirubin), and kidney functions (Blood urea nitrogen (BUN) and serum creatinine) will be evaluated.

Pan cultures (blood with/without wound culture, throat swab or sputum culture and urinary analysis and culture), will be withdrawn for baseline readings and redrawn if any signs of systemic inflammatory response,

ELIGIBILITY:
Inclusion Criteria:

All burn patients 1 to 5 years old with 10% or greater burn area of TBSA .

Exclusion Criteria:

* Patients with septic shock (evidence of infection and inotropes) .
* Burns more than 48 hours duration.

Ages: 1 Year to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2021-10-10 (Actual); Primary Completion 2022-07-16 (Actual); Study Completion 2022-07-16 (Actual)

PRIMARY OUTCOMES:
Incidence of sepsis during ICU stay will be recorded. | Through out study completion, average 30 days.
  Sepsis is defined by clinical criteria (temperature more than 38.9 °C, leukocytosis, thrombocytopenia, glucose intolerance, and/or new onset of ileus) and/or the presence of a positive blood culture in association with clinical signs of infection/sepsis. An increase in Procalcitonin level will be also used as an early laboratory marker for sepsis.

SECONDARY OUTCOMES:
Incidence of septic shock | Through out study completion, average 30 days.
  Defined by evidence of sepsis as previously mentioned and need for inotropes to support circulation.
Number of septic episodes | Throughout the study completion average 30 days.
  Sepsis is defined by clinical criteria (temperature more than 38.9 °C, leukocytosis, thrombocytopenia, glucose intolerance, and/or new onset of ileus) and/or the presence of a positive blood culture in association with clinical signs of infection/sepsis.
Length of stay | Through out study completion, average 30 day.
  days
PEdiatric Logistic Organ Dysfunction score 2 (PELOD-2) | Through out study completion, average 30 days
  Clinical assessment score used as diagnostic and prognostic tool of sepsis in pediatrics.It includes cardiovascular, neurologic, respiratory, hematologic, renal dysfunctions assessment adjusted to age.A higher PELOD-2 score correlates with a higher number of organ failures and mortality rate incidence.Each measurement gives a score form 0 to 6 and total score is directly proportional to increased morbidity and mortality probability.
Mortality rate | 30 days
  Number of patients
Days of mechanical ventilation | From date of randomization until the date of first documented progression or date of death from any cause,
  days

OTHER OUTCOMES:
serum Procalcitonin | Day 1 ,Day3 ,and on each incidence of sepsis, and through out study completion, average 30 days .
  ng/mL
serum IgG | Day 1 and Day 7.
  g/L.
serum C-reactive protein | Day 1 , and on each incidence of sepsis, assessed up to 30 days.
  mg/L.
Serum Malondialdehyde level (MDA) | Day 1 and Day 3
  nmol./ml
Serum Glutathione peroxidase level | Day 1 and Day 3
  U/L
Serum Micro RNA 25 | Day 1 and Day 3
  Fold change
Serum lactate | daily,through out study completion, average 30 days
  mmol/L
Demographic data as Age | Baseline
  In years.
Demographic data as Sex | Baseline
  sex of the study candidate.
Demographic data as total body surface area | Baseline
  Total body surface area
Depth of burn injured area | Baseline
  Rule of nine .,percentage of burn .
Hemodynamic data as heart rate | Through out study completion, average 30 days
  Heart rate in beats per minute
Hemodynamic data as oxygen saturation | Through out study completion, average 30 days
  oxygen saturation in percent
Hemodynamic data as body temperature. | Through out study completion, average 30 days
  body temperature in degrees Celsius
Hemodynamic data as Capillary refill time | Daily,through out study completion, average 30 days
  seconds
Hemodynamic data as systolic ,diastolic and mean non invasive blood pressure. | Through out study completion, average 30 days
  Systolic ,Diastolic and mean non invasive blood pressure in mmHg.

CONTACTS AND LOCATIONS:
Overall Officials: Hanan Mostafa, Principal Investigator — lecturer
Locations (1):
- Cairo University, Cairo, Egypt

REFERENCES:
- [Result] Galal NM. Pattern of intravenous immunoglobulins (IVIG) use in a pediatric intensive care facility in a resource limited setting. Afr Health Sci. 2013 Jun;13(2):261-5. doi: 10.4314/ahs.v13i2.9. PMID 24235922
- [Result] Lyons JM, Davis C, Rieman MT, Kopcha R, Phan H, Greenhalgh D, Palmieri T, Kagan R. Prophylactic intravenous immune globulin and polymixin B decrease the incidence of septic episodes and hospital length of stay in severely burned children. J Burn Care Res. 2006 Nov-Dec;27(6):813-8. doi: 10.1097/01.BCR.0000245421.54312.36. PMID 17091076
- [Result] Munster AM, Hoagland HC, Pruitt BA Jr. The effect of thermal injury on serum immunoglobulins. Ann Surg. 1970 Dec;172(6):965-9. doi: 10.1097/00000658-197012000-00006. No abstract available. PMID 5496482